CLINICAL TRIAL: NCT00504374
Title: Gene Polymorphisms and Symptoms in Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2006-0273; CA109043 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Epidemiology; Symptoms; Gene Polymorphisms; Questionnaire; Survey
MeSH Terms: conditions — Lung Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Leftover blood sample to look at certain genes in your blood that may affect your symptoms. If you did not have blood collected in the previous lung cancer study, you will have a blood sample (one tablespoon) drawn when you first agree to participate in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptoms Questionnaire: Patients with lung cancer.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Symptoms questionnaire lasting about 5 to 10 minutes.
  Other Names: Survey

SUMMARY:
Primary Objectives:

* Construct a prospective cohort of patients diagnosed with lung cancer and dispositioned for treatment and collect information on symptoms and symptom treatments at baseline and on follow-up.
* Develop preliminary statistical models incorporating genetic data (which will be obtained from an existing protocol, CPN 91-001, Margaret Spitz), disease-related variables (e.g., stage of disease, location of tumor), clinical health status (e.g., performance status, comorbid conditions), and sociodemographic characteristics (e.g., age, sex, race) for predicting the risk of severe and persistent symptoms.

Analytical aim: To determine if symptoms (e.g., fatigue, depression, lack of appetite) will differ in severity by IL-6 gene polymorphisms (-174G/C, -597G/A, -572G/C, -373An/Tn).

This study (NIH-CA109043, Reyes-Gibby, 2004-2009) builds upon an NIH-funded (NIH-CA55769, Spitz, 2003-2008) study of the molecular epidemiology of lung cancer.

DETAILED DESCRIPTION:
If you agree to take part in this study, upon being admitted for treatment, you will be asked about your symptoms (how severe they are and to what degree they affect your day-to-day functioning).

You will be asked to fill out a symptoms questionnaire each time you are at the clinic for your treatment and for your follow-up visits. The questionnaire will take about 5 to 10 minutes to complete each time.

You may also be contacted at home so that researchers can follow-up on your experience with symptoms (only if you are not able to come to the clinic for your chemoradiation treatment or follow-up visits). If you are contacted by phone, the call should last about 5 to 10 minutes each time.

Researchers will also try to collect some of your leftover blood (that was already drawn and stored for research studies) from a previous lung cancer study (Ecogenetics of Lung Cancer) that you participated in at M. D. Anderson. Researchers will use your leftover blood sample to look at certain genes in your blood that may affect your symptoms. If you did not have blood collected in the previous lung cancer study, you will have a blood sample (one tablespoon) drawn when you first agree to participate in this study.

This is an investigational study. Up to 320 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patient has lung cancer and is being treated at M. D. Anderson.
* At least 18 years of age
* Currently living in the United States
* Enrolled in CPN 91-001 (Molecular epidemiology of lung cancer)
* English or Spanish speaking

Exclusion Criteria:

* Patient is unable to understand the intent of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2006-06-13 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Patient Symptom Severity (MD Anderson Symptom Inventory Questionnaire) | Baseline (before), during (every week for 6 weeks), and after chemoradiation therapy (at 6-12 week intervals)

CONTACTS AND LOCATIONS:
Overall Officials: Cielito C. Reyes-Gibby, DrPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org